CLINICAL TRIAL: NCT01381991
Title: A Prospective Randomized Controlled Trial of the Efficacy of i-Scan for Detecting Reflux Esophagitis
Brief Title: The Efficacy of i-Scan for Detecting Reflux Esophagitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konkuk University Hospital (Other)
Responsible Party: Sung Noh Hong, M.D., Department of Internal Medicine, Konkuk University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: KUMCHSN03
Record Dates: First submitted 2011-05-17; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Gastroesophageal Reflux Disease; Reflux Esophagitis
Keywords: Gastroesophageal Reflux Disease; Reflux esophagitis; i-scan
MeSH Terms: conditions — Gastroesophageal Reflux; Esophagitis, Peptic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- i-scan-EGD (Experimental): Examination of GE junction using conventional WL as well as i-scan mode
  Interventions: Device: i-scan

INTERVENTIONS:
Device: i-scan — For all the study procedures, Pentax EPKi processor and high-resolution adult video endoscopes (EG-2890i; Pentax, Japan) with push button switch from WL to i-scan were used. I-scan consist of three modes of image enhancement including SE, CE, ant TE. For SE and CE, switching among three enhancement levels (2+,3+,4+) is possible. Although SE and CE modes can allow detailed observation of subtle mucosal irregularities, noise increases as enhancement becomes more intense. In addition, TE is possible to switch p (pit pattern), v (vessel), b (Barrett), e (esophagus), g (stomach) and c (colo-rectum) mode.
  Other Names: Pentax EPKi processor and EG-2890i endoscopy

SUMMARY:
Endoscopy is a widely used modality for the diagnosis and classification of Gastroesophageal reflux disease (GERD), and the extent of esophageal mucosal breaks on endoscopy can be assessed. However, there were some limitation in diagnosis of GERD using endoscopy

1. More than half of patients with GERD reveal no visible abnormality on conventional endoscopy, it is possible that minute mucosal changes are underestimated by conventional endoscopy due to the limitation of visual ability
2. In addition of uncertainty in detecting mucosal breaks, uncertainty in describing severity of mucosal injury can lead to inconsistency among interpreters. Interobserver agreement regarding diagnosis and classification of GERD using endoscopy is unsatisfactory to apply daily practice.

Thus, the development of a new method to define the intra-esophageal injury for use in daily practice is a worthwhile endeavor and developed, such as narrow-band imaging (NBI), Fuji Intelligent Chromoen-doscopy (FICE) and i-scan.

Among them, i-scan technology is the most recently developed image enhancing technology, which consists of three modes of image enhancement, i.e. surface enhancement (SE), contrast enhancement (CE), and tone enhancement (TE).

Thus, the investigators examined the hypothesis that i-scan can improve the detection rate of reflux esophagitis and inter-observer agreement between endoscopists compared with conventional white light (WL) endoscopic examination.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) is a condition that develops when reflux of stomach contents causes troublesome symptoms and/or complications. It is the most frequent problem in upper gastrointestinal tract in outpatient clinic and contributes substantially to morbidity and to costs. Endoscopy is a widely used modality for the diagnosis and classification of GERD, and the extent of esophageal mucosal breaks on endoscopy can be assessed. However, because more than half of patients with GERD reveal no visible abnormality on conventional endoscopy, it is possible that minute mucosal changes are underestimated by conventional endoscopy due to the limitation of visual ability.

In addition of uncertainty in detecting mucosal breaks, uncertainty in describing severity of mucosal injury can lead to inconsistency among interpreters. Asian gastroenterologists tend to diagnose endoscopically before they treat patients with symptoms suggestive of GERD and use the modified Los Angeles (LA) classification system that includes minimal changes as constituting a distinct grade of reflux esophagitis. In modified LA system, minimal change esophagitis is characterized by the mucosa such as erythema and/or whitish turbidity. However, because substantial overlap is noted between normal and minimal change, minimal change and LA class A, and LA class A and B, interobserver agreement regarding diagnosis and classification of reflux esophagitis is unsatisfactory to apply daily practice. Thus, the development of a new method to define the intra-esophageal injury for use in daily practice is a worthwhile endeavor.

Currently, new imaging technologies have applied in endoscopy to improve detecting and differentiating the subtle mucosal changes using digital contrast method such as narrow-band imaging (NBI), Fuji Intelligent Chromoen-doscopy (FICE) and i-scan. Among them, i-scan technology is the most recently developed image enhancing technology, which consists of three modes of image enhancement, i.e. surface enhancement (SE), contrast enhancement (CE), and tone enhancement (TE). SE enhances light-dark contrast and CE adds blue color in relatively dark areas digitally, by obtaining luminance intensity data for each pixel. Applying SE and CE might allow detailed observation of subtle irregularities around the surface and TE analyzes the individual RGB components of a normal image and recombines the color frequencies of each component to enhance minute mucosal structures with subtle color changes.

Thus, the investigators examined the hypothesis that i-scan can improve the detection rate of reflux esophagitis and inter-observer agreement between endoscopists compared with conventional white light (WL) endoscopic examination

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 80 years
* completed standard questionnaire including upper gastrointestinal symptoms
* underwent screening endoscopy

Exclusion Criteria:

* a patients with history of gastrointestinal surgery such as gastrectomy, fundoplication, or distal esophagectomy
* a patients were not able to record video clips during the period of examination of the gastro-esophageal junction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2010-07; Primary Completion 2010-11 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To compare reflux esophagitis detection rate | from 2 to 3months after completeion of patients' enrollement
  using videoclip (for endoscopic finding of GE junction) of WL-EGD vs. i-scan-EGD of all enrolled patients

SECONDARY OUTCOMES:
To evaluate the interobserver agreement using modified LA classification | from 3 to 4 months after completeion of patients' enrollement
  using videoclip (for endoscopic finding of GE junction) of WL-EGD vs. i-scan-EGD from 60 randomly selected enrolled patients

CONTACTS AND LOCATIONS:
Overall Officials: Sung Noh Hong, M.D., Principal Investigator — Konkuk University Medical Center,Konkuk University School of Medicine
Locations (1):
- Healthcare Center, Digestive Disease Center, Konkuk University Medical Center, Seoul, South Korea